CLINICAL TRIAL: NCT00675649
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Parallel-group Study Evaluating the Efficacy and Safety of Golimumab Administered Subcutaneously in Symptomatic Subjects With Severe, Persistent Asthma
Brief Title: A Clinical Trial Evaluating the Safety and Effectiveness of Golimumab in Patients With Severe, Persistent Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014980; C0524T26; EudraCT No.: 2007-005699-15
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Injections; Severe, persistent asthma
MeSH Terms: conditions — Asthma | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental)
  Interventions: Biological: CNTO 148 / Golimumab
- 002 (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: CNTO 148 / Golimumab — 100 mg sc injection every 4 weeks from week 0 to week 20
  Arms: 001
Biological: placebo — placebo sc injection every 4 weeks from week 0 to week 20
  Arms: 002

SUMMARY:
The purpose of this study is to assess the safety and effects (good and bad) of golimumab therapy in patients with severe, persistent asthma.

DETAILED DESCRIPTION:
Golimumab is a type of tumor necrosis factor (TNF) inhibitor. TNF is a naturally occurring substance in the body and this substance may cause long-term inflammation. Golimumab may help treat this disease by blocking the activity of TNF in the body and reducing the symptoms of severe, persistent asthma.This study will assess the safety and effectiveness of subcutaneously (under the skin) administered golimumab and determine if there is a reduction of signs and symptoms in patients with active severe, persistent asthma. The effect of subcutaneously (SC) administered golimumab on the quality of life in patients with severe, persistent asthma will also be assessed. About 200 patients will take part in the study at approximately 60 centers worldwide. Participation in the study will last for about 42 weeks. The study consists of 3 phases: the screening phase (lasting between 1 and 4 weeks), the treatment phase (20 weeks), and the follow-up phase (20 weeks). Visits are scheduled to occur once every 4 weeks during the treatment and follow-up phases of the study. Patients eligible to take part in this study will be randomly placed into one of the following study groups: Group 1: Placebo (an inactive or dummy treatment that looks the same as the study drug, golimumab, but does not contain any active medication) from Week 0 through Week 20. Group 2: Golimumab 100 mg from Week 0 through Week 20. This study is "blinded." This means that neither patient nor study doctor will know in which group a patient is placed. However, if needed for safety or health reasons, the study doctor can find out a patient's study group at any time.

Patients will receive an injection (under the skin) of placebo (Group 1) or golimumab 100 mg (Group 2) every 4 weeks from Week 0 through Week 20.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma for >= 3 years and a diagnosis of severe, persistent asthma for >= 1 year prior to screening
* Reversible airway obstruction
* Continuous treatment with high dose inhaled corticosteroids and long-acting Beta2-agonist for at least 3 months prior to screening
* At least 1 occasion in the previous 6 months when worsening of asthma required treatment with additional steroids (intravenous or oral)
* Score of >= 2 points on the Asthma Control Questionnaire (ACQ) at screening

Exclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD), cystic fibrosis, or other significant respiratory disorder
* Life-threatening asthma attack requiring intubation in the 6-month period prior to screening
* Steroid use at a dose > 20 mg of prednisone at the screening visit
* Known malignancy or history of malignancy
* Previous exposure to anti-TNF therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05

PRIMARY OUTCOMES:
The primary endpoint is the time to first severe asthma exacerbation through Week 24. | Week 24

SECONDARY OUTCOMES:
Secondary endpoints include the number of severe asthma exacerbations through Week 24, number of clinically significant asthma exacerbations through Week 24, and change from baseline in Asthma Quality of Life Questionnaire (AQLQ) overall score at Week 24 | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.